CLINICAL TRIAL: NCT05328700
Title: Effectiveness of Neuromuscular Kinesiology Taping in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNM_CC
Record Dates: First submitted 2022-03-22; First posted 2022-04-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Fasciitis, Plantar
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Experimental)
  Interventions: Other: Kinesiotaping
- Tape (Placebo Comparator)
  Interventions: Other: Tape

INTERVENTIONS:
Other: Kinesiotaping — Perform a neuromuscular bandage with kinesiotape in patients with plantar fasciitis
  Arms: kinesiotaping
Other: Tape — Perform a neuromuscular bandage with tape (Hipofix(R)) in patients with plantar fasciitis
  Arms: Tape

SUMMARY:
One of the pathologies most studied and treated with kinesiotape (KT) is plantar fasciitis (PF). In most of the studies reviewed, it is concluded that there is an improvement in the symptoms of PF when treated with KT: either combined with other therapies or as a single treatment compared to placebo. However, most current studies have limitations because the sample is small, the effect size is small, and the evidence is insufficient or of low quality.

In the present work, the aim is to study the effectiveness of KT in PF, and to compare the results with those obtained in a placebo group, which is treated with tape. The researchers will assess the decrease in symptoms prior to performing other definitive treatments. In addition, the variability of the painful symptoms and the durability of the bandage will be studied, in order to determine whether it can be used in the short or long period of time, being able to take it into account and supposing a supplement to the pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* People with acute plantar fasciitis with less than 3 months of evolution
* Who present pain in the fascia both during ambulation and on palpation
* Ecographic image compatible with plantar fasciitis (> 4 mm)
* The condition has not be previously treated with other treatment

Exclusion Criteria:

* Condition with no sintomatology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of Pain | Change from baseline (before intervention) to one day, two days, three days and four days after intervention
  A visual analogue scale of pain will assess from 0, no pain, to 10, the worst possible pain

SECONDARY OUTCOMES:
Bandage durability | Change from baseline (the bandage is put on) until the first day that the loss of the bandage is documented, assessed up to 7 days
  Period of time in days from when the bandage is put on until it comes off

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de València, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided